CLINICAL TRIAL: NCT04875325
Title: Recurrent Disease Detection After Resection of Pancreatic Adenocarcinoma Using a Standardized Surveillance Strategy: a Nationwide Randomized Controlled Trial
Brief Title: Recurrent Disease Detection After Resection of Pancreatic Adenocarcinoma Using a Standardized Surveillance Strategy
Acronym: RADAR-PANC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Pancreatic Cancer Group (DPCG) (Unknown); University of Birmingham (Other)
Responsible Party: Principal Investigator, Prof. dr. I.Q. Molenaar, MD, PhD, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL67115.041.18; 20-762 (Other: METC Utrecht)
Record Dates: First submitted 2021-03-17; First posted 2021-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma; Recurrent Pancreatic Ductal Adenocarcinoma
Keywords: Standardized Surveillance; Follow-up; CA 19-9; Computed Tomography Scan

STUDY DESIGN:
Intervention Model Description: Trials within Cohorts (TwiCs)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized surveillance (Experimental): Standardized surveillance strategy with routine imaging and serum tumor marker testing.
  Interventions: Other: Standardized surveillance
- Non-standardized surveillance (No Intervention): Non-standardized surveillance strategy according to current clinical practice.

INTERVENTIONS:
Other: Standardized surveillance — Standardized 3-monthly surveillance with routine imaging and serum tumor marker testing.
  Arms: Standardized surveillance

SUMMARY:
A randomized controlled trial, nested within an existing prospective cohort (Dutch Pancreatic Cancer Project; PACAP) and the United Kingdom (UK) Pancreas Cancer: Observations of Practice and survival; PACOPS) according to the 'trials within cohorts' (TwiCs) design in which the effect of a standardized surveillance, with serial tumor marker testing and routine imaging, compared to current non-standardized practice, on overall survival and quality of life in patients with primary resected PDAC is investigated. The most important secondary endpoint is quality of life. Other secondary endpoints are clinical and radiological patterns of PDAC recurrence, the compliance of patients to our standardized follow-up strategy, the impact of a standardized surveillance on (eligibility for) additional treatment, and the tolerance of additional treatment. The need for this clinical trial is emphasized by the the emergence of more potent local and more effective systemic treatments for PDAC recurrence, leading to a rising interest in early diagnosis by a standardized approach to follow-up with routine imaging and serial serum tumor marker testing.

DETAILED DESCRIPTION:
Rationale: Radical resection combined with (neo)adjuvant chemotherapy offers the best chances for long-term survival for patients with resectable localized pancreatic ductal adenocarcinoma (PDAC). However, even after radical resection, almost all patients will experience local and/or distant disease recurrence after sufficient follow-up, mostly within 2 years. There is a lack of evidence based effective therapeutic options for the significant group of patients with local recurrence only, in terms of improved survival and/or quality of life. In the case of metastatic disease effective chemotherapy has shown to improve survival, but with a median gain survival of 3-4 months. Taken together, this had led to a hesitant attitude towards postoperative recurrence-focused follow-up. Therefore, in most European countries, including the Netherlands, a standardized approach to follow-up after surgery for PDAC is lacking. Furthermore, current PDAC guidelines regarding follow-up are based on expert opinion and other low-level evidence. However, the emergence of more potent local and more effective systemic treatments for PDAC has led to a rising interest in early diagnosis of PDAC recurrence. To detect PDAC recurrence at an early stage and identify patients with good performance status who are most likely to benefit from additional (experimental) treatment, a standardized approach to follow-up with routine imaging and serial serum tumor marker testing is needed. To determine whether early detection of recurrence can lead to improved survival and quality of life, further studies are warranted.

Objective: The main objective is to evaluate the impact of a standardized surveillance, with serial tumor marker testing and routine imaging, on overall survival and quality of life in patients with primary resected PDAC, compared to current non-standardized practice.

Study design: A randomized controlled trial, nested within an existing prospective cohort (Dutch Pancreatic Cancer Project; PACAP) and the United Kingdom (UK) Pancreas Cancer: Observations of Practice and survival; PACOPS) according to the 'trials within cohorts' (TwiCs) design.

Study population: PACAP or PACOPS-participants with histologically confirmed radical resection (R0-R1) of PDAC, who provided informed consent for being randomized in future studies.

Interventions: Standardized surveillance, existing of clinical evaluation, serum cancer antigen (CA) 19-9 testing, and contrast-enhanced computed tomography (CT-) imaging of chest and abdomen every 3 months during the first 2 years after surgery.

Comparison: Non-standardized clinical follow-up.

Endpoints: The main study endpoint is overall survival. The most important secondary endpoint is quality of life. Other secondary endpoints are clinical and radiological patterns of PDAC recurrence, the compliance of patients to our standardized follow-up strategy, the impact of a standardized surveillance on (eligibility for) additional treatment, and the tolerance of additional treatment.

ELIGIBILITY:
Inclusion criteria:

* Participation in the PACAP and PACOPS-cohort with written informed consent for being randomized in future studies
* Histologically confirmed macroscopically radical resected (R0-R1) pancreatic adenocarcinoma
* Minimum age of 18 years

Exclusion Criteria:

* Exclusion criteria for contrast-enhanced CT-scan, following the protocol of the department of radiology in each affiliated hospital
* Mentally or physically incapable of consent
* Participation in other studies with a study-specific follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of PDAC resection until date of death from any cause or date of last follow-up, whichever came first, assessed up to 24 months
  The interval between the date of PDAC resection and either death from any cause or last follow-up.

SECONDARY OUTCOMES:
Compliance of the standardized surveillance strategy | Through completion of patient inclusion, an average of 1.5 years
  The percentage of patients that either accepts or refuses participation in the intervention-arm, i.e. is willing to undergo a standardized follow-up regime.
Recurrence-free interval | From date of PDAC resection until date of first radiological signs of recurrence, or last follow-up if recurrence is not observed, whichever came first, assessed up to 24 months
  The interval between the date of PDAC resection and the date of first radiological signs of recurrence, or last follow-up if recurrence is not observed.
Prognostic patient specific characteristics and tumor related factors for disease recurrence | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months
Role of serum tumor marker testing in detecting recurrent PDAC assessed by the calculated diagnostic accuracy values | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months
Eligibility for additional (experimental) treatment at the time of recurrence diagnosis based on the ECOG or Karnofsky performance state, or inclusion criteria for study-related treatment of recurrence | At the time of recurrence diagnosis. Assessed through the study, up to 24 months
Reasons to refrain from treatment for recurrence | At the time the patient is assessed eligible for additional treatment. Assessed through the study, up to 24 months
  e.g. poor condition, patients wish, deteriorated condition, progressive disease, advise treating clinician, death, wait-and-see, age.
Patients' tolerance of additional treatment for PDAC recurrence as assessed by incidence of adverse events (graded according to NCI CTCAE Version 5.0) | Through study completion, an average of 2 years
Morbidity associated with diagnostic testing assessed by the side-effects of diagnostic testing (i.e. fear of disease recurrence) | From date of randomization until disease recurrence or last follow-up, whichever came first, assessed up to 24 months
Patient reported non-disease specific health-related Quality of Life (HRQoL) as assessed using the EQ-5D-5L | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Overall costs of a standardized surveillance strategy versus the costs as incurred with the current non-standardized follow-up assessed according to the EQ-5D questionnaire as part of the PACAP and PACOPS-project, and calculated using to a Markov model | After study completion (estimated duration of 3.5 years)
Patient reported chemotherapy-induced peripheral neuropathy as assessed using the EORTC QLQ-CIPN20 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Patient reported Quality of Life as assessed using the happiness, hospital, anxiety and depression scale (HADS) | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Patient reported Quality of Life as assessed using Exocrine Pancreatic Insufficiency (EPI) questionnaire | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Patient reported Quality of Life as assessed using the worry of progression of cancer scale (WOPS) | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Patient reported cancer-specific HRQoL as assessed using the EORTC QLQ-C30 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.
Patient reported tumor-specific HRQoL as assessed using the EORTC LQPAN26 | At baseline and at 3, 6, 9, 12, 18 and 24 months and every subsequent year after enrollment in the PACAP and PACOPS-cohort. Assessed through study completion, up to 24 months
  Part of the Patient Reported Outcome Measures (PROMs) that are being standardly measured in PACAP and PACOPS-participants.

OTHER OUTCOMES:
Clinical patterns of disease recurrence assessed by the patients symptoms as reported in the electronic patient dossier: explanatory | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months
Clinical patterns of disease recurrence assessed by physicial examination as reported in the electronic patient dossier: explanatory | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months
Clinical patterns of disease recurrence assessed by blood test results as reported in the electronic patient dossier: explanatory | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months
Radiological patterns of disease recurrence assessed by information from imaging reports from the electronic patient dossier: explanatory | From date of randomization until disease recurrence or last follow-up, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: I. Q. Molenaar, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); H. C. van Santvoort, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU); M. G.H. Besselink, MD, PhD, Principal Investigator — Academic Medical Center - Cancer Center Amsterdam; L. A. Daamen, MD, PhD, Principal Investigator — Regional Academic Cancer Center Utrecht (RACU)
Locations (11):
- Netherlands (10):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht UMC, Maastricht, Limburg
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Amsterdam University Medical Center VUmc, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Amsterdam University Medical Center AMC, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Sint Antonius Ziekenhuis, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht, Utrecht
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data generated during the RADAR-PANC trial will be made available to other researcher upon request from I.Q. Molenaar.
Supporting Information: Study Protocol
Access Criteria: Upon request.

REFERENCES:
- [Derived] Daamen LA, van Goor IWJM, Groot VP, Andel PCM, Brosens LAA, Busch OR, Cirkel GA, Mohammad NH, Heerkens HD, de Hingh IHJT, Hoogwater F, van Laarhoven HWM, Los M, Meijer GJ, de Meijer VE, Pande R, Roberts KJ, Stoker J, Stommel MWJ, van Tienhoven G, Verdonk RC, Verkooijen HM, Wessels FJ, Wilmink JW, Besselink MG, van Santvoort HC, Intven MPW, Molenaar IQ; Dutch Pancreatic Cancer Group. Recurrent disease detection after resection of pancreatic ductal adenocarcinoma using a recurrence-focused surveillance strategy (RADAR-PANC): protocol of an international randomized controlled trial according to the Trials within Cohorts design. Trials. 2024 Jun 20;25(1):401. doi: 10.1186/s13063-024-08223-5. PMID 38902836